CLINICAL TRIAL: NCT05536570
Title: Management of Functional Thoracic Outlet Syndrome (TOS - Whiplash) With IncobotulinumtoxinA Injections
Brief Title: Whiplash-induced Thoracic Outlet Syndrome Treated With Botulinum Toxin.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King, David, MD (Individual)
Collaborators: MERZ PHARMA (Unknown)
Responsible Party: Principal Investigator, David King, Neurologist, Principal Investigator, Assistant Professor of Medicine, King, David, MD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMSI-1
Record Dates: First submitted 2022-07-27; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Thoracic Outlet Syndrome; Whiplash Injuries
MeSH Terms: conditions — Thoracic Outlet Syndrome; Whiplash Injuries

STUDY DESIGN:
Intervention Model Description: Patients who have neck pain and arm paresthesia following a side-on collision
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: IncobotulinumtoxinA 100 UNT — Scalene injection

SUMMARY:
Whiplash injuries following car accident are common, it has been reported to affect 83% of individuals injured in traffic collisions (Yadla S, 2007). The condition is caused by a rapid acceleration followed immediately by a rapid deceleration of the neck and head. The annual North American incidence rate is estimated to be 600 per 100,000 people (Holm LW, 2008). The condition is costly for society and disabling/painful for the patients. Depending on the collision type, the biomechanics of muscles will be affected differently and consequently the clinical presentation will vary. T-bone type of car collisions (when the front of one vehicle strikes the side of another) may induce thoracic outlet syndrome (TOS) following compression on the nerve and artery bundle by the scalene muscles (lateral stabilizers of the neck). An appropriate and detailed examination of the patient is necessary to identify the cause of the resulting pain and disability. Once a functional thoracic outlet syndrome is identified the proposal is to treat this with botulinum toxin.

DETAILED DESCRIPTION:
TOS symptoms will typical emerge within 24-48 hours following the accident. The duration will depend on the level of severity of the muscle damage. If the severity is a grade 1 (mild damage to individual muscle fibers), symptoms may last up to 3 weeks. If the severity is a grade 2 (more extensive damage with more muscle fibers involved/no complete rupture), symptoms may last up to 3 months. However, in many cases, due to muscle swelling and consequently compression of the nerve plexus, a persistent reflex spasm of muscle develops.

A potentially effective treatment strategy, in patients presenting TOS associated clinical symptoms in the proper distribution, is to relax the scalene muscles that surround the nerve plexus. Botulinum toxin, such as incobotulinumtoxinA (XEOMIN, Merz herapeutics), have been shown to be effective and safe in relaxing these muscles in conditions like spasticity, blepharospasm and cervical dystonia (Kanovský P, 2009; Benecke R, 2005; Roggenkämper P, 2005). It is hypothesised that a subtype of whiplash defined as functional TOS could be improved with incobotulinumtoxinA injections into the medial scalene muscle. IncobotulinumtoxinA when injected into the medial scalene is expected to induce muscle relaxation which leads to nerve plexus decompression. The effect is anticipated to last approximately 3 months, which is the duration of effect of botulinum toxins type A. A similar effect can be induced using a local anaesthetic, such xylocaine, since it has a similar mechanism of action, but his effect should be short lived.

ELIGIBILITY:
Inclusion Criteria:

* • Patient must have been diagnosed with a muscle strain to the lateral neck muscles following a car accident and there must be the following clinical signs of TOS: pain in the proper distribution, weakened grip, shoulder elevation on the appropriate side and numbness or tingling in the arm or fingers;

  * Patient must have no signs suggesting a radiculopathy that could account for similar symptoms;
  * Patient must have a PDQ >70, i.e. in the moderate to very severe disability range;
  * Patient must experience symptoms for longer than 3 months;
  * Patient must have had the accident leading to whiplash within the last 3 years;
  * Patient must be 18 years of age or older;
  * Patient must be eligible and agreeable to treatment with BoNT-A;
  * Patient must be toxin-naïve for the treatment of the cervical region, or have undergone a six months washout period;
  * Patient must be English speaking;
  * Patient must be able to provide informed consent.

Exclusion Criteria:

* • Patient unable or unwilling to complete the necessary assessment tasks;

  * Patient with hypersensitivity to botulinum neurotoxin type A or to any of the excipients, generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert-Eaton syndrome), or infection or inflammation at the proposed injection site(s);
  * Patient who requires physiotherapy and/or massage therapy;
  * Patient for whom concomitant medications are not controlled at study start and/or may require change/adjustment during the study;
  * Patient who had surgery which may interfere with the study;
  * Women who are pregnant or nursing, or women in age of reproduction not using a contraceptive method;
  * Patient in active litigation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain disability as assessed using the PDQ at Week 4. | week 4
  PDQ before and after treatment. Pain Disability Questionnaire (Guides to the Evaluation of Permanent Impairment, Sixth Edition.
  0= No pain related impairment 1-70= Mild pain related impairment 71-100=Moderate pain related impairment 101-130= Severe pain related impairment 131-150= Extreme pain related impairment

SECONDARY OUTCOMES:
Shoulder Elevation | week 4
  Change from baseline in shoulder elevation as assessed by measurement on photograph (clavicular angle) at Weeks 4, 12 and 16;
Grip Strength | Week 4
  3. Change from baseline in grip strength as assessed using a dynamometer at Weeks 4, 12 and 16;
Pinch Test | WFeek 4
  4. Change from baseline in fine motor test (pinch test) at Weeks 4, 12 and 16;

CONTACTS AND LOCATIONS:
Locations (1):
- Private Office, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No